CLINICAL TRIAL: NCT00579657
Title: Effects of High Protein and High Cereal Fiber Diets on Insulin Sensitivity in Overweight and Obese Subjects With the Metabolic Syndrome - The PROFIMET Study
Brief Title: Protein, Fiber, and Metabolic Syndrome - The PROFIMET Study
Acronym: PROFIMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Medical University of Vienna (Other); Heinrich-Heine University, Duesseldorf (Other); University Hospital Tuebingen (Other); Charite University, Berlin, Germany (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Coventry University (Other)
Responsible Party: Principal Investigator, Prof Weickert, Martin O., MD, FRCP, Study PI, University Hospitals Coventry and Warwickshire NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: mow_PROFIMET; BMBF Profimet 0313826A
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Overweight; Obesity; Metabolic Syndrome
Keywords: parameters of metabolic syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome | interventions — Diet, High-Protein; Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Intervention: 'control diet, supported by dietary supplement twice daily'
  control diet [carbohydrates 55(50 - 60)% , protein 15(10 - 20)% protein; fat ca. 30% of energy content; dietary fiber < 15 g/1000 kcal and day; intensive dietary advice plus supplement (2 x basic supplement daily)]
  Interventions: Other: control diet, supported by dietary supplement twice daily
- 2 (Experimental): Intervention: 'high cereal fiber diet, supported by dietary supplement twice daily'.
  high cereal fiber diet [carbohydrates 55(50 - 60)% , protein 15(10 - 20)% protein; fat ca. 30% of energy content; dietary fiber > 20 g/1000 kcal and day; intensive dietary advice plus supplement (2 x basic supplement including 2 x 15 g cereal fiber daily)]
  Interventions: Other: high cereal fiber diet, supported by dietary supplement twice daily
- 3 (Experimental): Intervention: 'high protein diet, supported by dietary supplement twice daily'
  high protein diet [carbohydrates 40 - 45% , protein > 25 - 30%; fat ca. 30% of energy content; dietary fiber < 15 g/1000 kcal and day; intensive dietary advice plus supplement (2 x basic supplement including 2 x 25 g whey and plant protein daily)]
  Interventions: Other: high protein diet, supported by dietary supplement twice daily
- 4 (Experimental): Intervention: "diet moderately high both in cereal fiber and protein, supported by dietary supplement twice daily".
  high cereal fiber/high protein (MIX) moderately high cereal fiber/high protein diet (carbohydrates 45- 50)% , protein 20 - 25%; fat ca. 30% of energy content; dietary fiber 15 - 20 g/1000 kcal and day; intensive dietary advice plus supplement (2 x basic supplement including 2 x 15 g cereal fiber and 2 x 25 g whey and plant protein daily)
  Interventions: Other: diet moderately high both in cereal fiber and protein, supported by dietary supplement twice daily

INTERVENTIONS:
Other: control diet, supported by dietary supplement twice daily — control diet, see above
  Arms: 1
Other: high cereal fiber diet, supported by dietary supplement twice daily — high cereal fiber diet, see above
  Arms: 2
Other: high protein diet, supported by dietary supplement twice daily — high protein diet, see above
  Arms: 3
Other: diet moderately high both in cereal fiber and protein, supported by dietary supplement twice daily — MIX diet, see above
  Arms: 4

SUMMARY:
Randomized controlled single-blinded intervention study in 111 overweight and obese subjects with risk factors of developing type 2 diabetes, with the aim to investigate effects of isoenergetic high cereal fiber as compared with high protein diets over 6 and 18 weeks.

Proof of principle study with analysis according to study protocol, investigating whether isoenergetic high cereal fiber and high protein diets with comparable fat contents, if adhered to and after exclusion of known confounders such as changes in body weight, intake of drugs with known effects on insulin sensitivity, or relevant changes in physical activity, indeed affect insulin sensitivity.

DETAILED DESCRIPTION:
This is a randomized controlled single-blinded intervention study in 111 overweight and obese subjects with risk factors of developing type 2 diabetes, with the aim to investigate effects of isoenergetic high cereal fiber versus high protein diets over 6 and 18 weeks. We also investigate effects of a combined high-cereal-fiber/high-protein (mix) diet, and effects in a control group. All diets are based on foods from plants and whey products commonly assumed to be healthy. This trial is designed as a proof of principle study focusing on participants that are likely to adhere to the respective isoenergetic diets, in order to show whether high protein versus high cereal fiber diets indeed affect insulin sensitivity, as indicated by epidemiological observations. Study participants will receive intensive and regular nutritional advice in order to achieve the respective dietary targets. Dietary adherence of the participants will be supported by providing tailored dietary supplements in all four groups, twice daily over 18 weeks. Supplements are provided for twice daily consumption for all participants in all four dietary intervention groups, throughout the 18-wk intervention (each of the participants will be instructed to consume a total 252 portions of tailored supplements during the intervention, which will handed to the participants in sealed single portions at weeks 0, 3, 6 and 12, totalling 63 portions at each occasion). The packaging of the sealed portions for the 4 intervention arms do not indicate the type of dietary intervention for the participant, but are coded for identification by the supplier. Energy contents of the supplements are considered when calculating individual energy intake. Supplements have been specifically designed for this intervention study, in order to facilitate achieving dietary targets. A 6 week strictly controlled isoenergetic study period (regular group and individual sessions, daily food diaries/FFQs over the first 6 weeks with adaptation of food intake, if necessary, as indicated by direct analysis of FFQs and food protocols, and by weighing the participants; 3-day food protocols at weeks 0, 6, 12, and 18; various biomarkers of dietary adherence) will be followed by a further 12 week ad libitum period, with ongoing intake of the respective diet including the supplements, but no further dietary advice. The primary outcome measure is the detection of diet-induced changes in insulin sensitivity during weight maintaining isoenergetic conditions. Secondary outcomes are changes in factors that may explain potential diet-induced alterations of insulin sensitivity. During the 12-weeks ad libitum period we will further investigate potential effects of the respective diet on changes in body weight, body composition and biomarkers related to energy intake. Participants will be re-invited for anthropometric measurements and measurement of biomarkers in blood (18 weeks after completion of the study), as well as for taking a second muscle tissue biopsy (subset of participants that agreed to this procedure).

ELIGIBILITY:
Inclusion Criteria:

* Waist > 80 cm (females) or > 94 cm (males)
* BMI > 25 kg/m²
* IFG, IGT, or insulin resistance; and/or dyslipidemia; and/or high blood pressure
* Willingness to comply with one of the randomly assigned diets over the study period

Exclusion Criteria:

* Diabetes type 1 and type 2
* Pregnancy
* Allergies including food allergies
* Metal implants
* Chronic disease of heart, kidney, or liver
* Relevant deviation of body weight during isoenergetic 6-weeks period (+/- 3 kg)
* Intake of drugs with known impact on whole-body insulin sensitivity during the study (e.g. cortisone, ASS, antibiotics)
* Missing data about primary outcome measures (Clamp data, data about dietary intake from food diaries or 3-day food protocols)
* Significant deviation from dietary targets during the monitored 6 weeks isoenergetic period (e.g. significant deviation from 30% target for dietary fat in all groups, intake of a low protein or low fiber diet in the high protein or high fiber groups, respectively)

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change in insulin sensitivity | 6 weeks
  whole-body insulin sensitivity measured with euglycemic hyperinsulinemic clamp; hepatic insulin sensitivity measured with stable isotope techniques (DD-glucose) during the clamps; relation with secondary outcome measures
change in insulin sensitivity | 18 weeks
  whole-body insulin sensitivity measured with euglycemic hyperinsulinemic clamp; hepatic insulin sensitivity measured with stable isotope techniques (DD-glucose) during the clamps; relation with secondary outcome measures

SECONDARY OUTCOMES:
factors that may contribute explaining changes in primary outcome measures | 0, 6, 18 weeks
  body fat composition (MRI and ADP), liver fat (H1-spectroscopy); hormones, adipokines, inflammatory and metabolic markers; insulin signaling pathways in adipose tissue (gene expression and protein level); changes in gut microbiota; bile acids; metabolite profiles; amino acid composition in diet and circulating blood. Relation of secondary outcome measures with primary outcome measures.
biomarkers indicating dietary adherence | 0, 6, 18 weeks
  urinary nitrogen/creatine ratio and fecal BCAA as markers for protein intake; fecal SCFA and breath hydrogen levels as markers for fermentable fiber intake; HDL cholesterol as marker for carbohydrate intake
development of indices for the prediction of insulin resistance (liver, whole-body) | baseline, validation after 6 -18 weeks
development for indices for the prediction of fat mass (liver, abdominal) | baseline, validation after 6 -18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Weickert, MD, Study Chair — University Hospitals Coventry & Warwickshire; and University of Warwick, UK; Andreas FH Pfeiffer, Prof, Study Director — German Institute of Human Nutrition Potsdam-Rehbrücke; Charité-University-Medicine Berlin
Locations (4):
- Germany (3):
  - Deutsches Diabetes Zentrum; Heinrich Heine University, Düsseldorf
  - Diagnostic and Interventional Radiology, Klinikum Ernst von Bergmann, Academic Teaching Hospital, Charité University Medicine Berlin, Potsdam
  - Eberhard-Karls University Tübingen, Section on Experimental Radiology, Department of Diagnostic and Interventional Radiology, Tübingen
- University Hospitals Coventry and Warwickshire NHS Trust, Coventry, Warwickshire, United Kingdom

REFERENCES:
- [Background] Gogebakan O, Kohl A, Osterhoff MA, van Baak MA, Jebb SA, Papadaki A, Martinez JA, Handjieva-Darlenska T, Hlavaty P, Weickert MO, Holst C, Saris WH, Astrup A, Pfeiffer AF; DiOGenes. Effects of weight loss and long-term weight maintenance with diets varying in protein and glycemic index on cardiovascular risk factors: the diet, obesity, and genes (DiOGenes) study: a randomized, controlled trial. Circulation. 2011 Dec 20;124(25):2829-38. doi: 10.1161/CIRCULATIONAHA.111.033274. Epub 2011 Nov 21. PMID 22104550
- [Background] Isken F, Klaus S, Osterhoff M, Pfeiffer AF, Weickert MO. Effects of long-term soluble vs. insoluble dietary fiber intake on high-fat diet-induced obesity in C57BL/6J mice. J Nutr Biochem. 2010 Apr;21(4):278-84. doi: 10.1016/j.jnutbio.2008.12.012. Epub 2009 Apr 14. PMID 19369060
- [Background] Weickert MO, Pfeiffer AF. Low-glycemic index vs high-cereal fiber diet in type 2 diabetes. JAMA. 2009 Apr 15;301(15):1538; author reply 1538-9. doi: 10.1001/jama.2009.483. No abstract available. PMID 19366767
- [Background] Weickert MO, Pfeiffer AF. Metabolic effects of dietary fiber consumption and prevention of diabetes. J Nutr. 2008 Mar;138(3):439-42. doi: 10.1093/jn/138.3.439. PMID 18287346
- [Background] Weickert MO, Mohlig M, Schofl C, Arafat AM, Otto B, Viehoff H, Koebnick C, Kohl A, Spranger J, Pfeiffer AF. Cereal fiber improves whole-body insulin sensitivity in overweight and obese women. Diabetes Care. 2006 Apr;29(4):775-80. doi: 10.2337/diacare.29.04.06.dc05-2374. PMID 16567814
- [Background] Weickert MO, Mohlig M, Koebnick C, Holst JJ, Namsolleck P, Ristow M, Osterhoff M, Rochlitz H, Rudovich N, Spranger J, Pfeiffer AF. Impact of cereal fibre on glucose-regulating factors. Diabetologia. 2005 Nov;48(11):2343-53. doi: 10.1007/s00125-005-1941-x. Epub 2005 Sep 20. PMID 16172868
- [Result] Weickert MO, Roden M, Isken F, Hoffmann D, Nowotny P, Osterhoff M, Blaut M, Alpert C, Gogebakan O, Bumke-Vogt C, Mueller F, Machann J, Barber TM, Petzke KJ, Hierholzer J, Hornemann S, Kruse M, Illner AK, Kohl A, Loeffelholz CV, Arafat AM, Mohlig M, Pfeiffer AF. Effects of supplemented isoenergetic diets differing in cereal fiber and protein content on insulin sensitivity in overweight humans. Am J Clin Nutr. 2011 Aug;94(2):459-71. doi: 10.3945/ajcn.110.004374. Epub 2011 Jun 1. PMID 21633074
- [Result] Weickert MO, Arafat AM, Blaut M, Alpert C, Becker N, Leupelt V, Rudovich N, Mohlig M, Pfeiffer AF. Changes in dominant groups of the gut microbiota do not explain cereal-fiber induced improvement of whole-body insulin sensitivity. Nutr Metab (Lond). 2011 Dec 17;8:90. doi: 10.1186/1743-7075-8-90. PMID 22177085
- [Result] Hattersley JG, Mohlig M, Roden M, Arafat AM, Loeffelholz CV, Nowotny P, Machann J, Hierholzer J, Osterhoff M, Khan M, Pfeiffer AF, Weickert MO. Quantifying the improvement of surrogate indices of hepatic insulin resistance using complex measurement techniques. PLoS One. 2012;7(6):e39029. doi: 10.1371/journal.pone.0039029. Epub 2012 Jun 22. PMID 22761721
- [Result] Weickert MO. What dietary modification best improves insulin sensitivity and why? Clin Endocrinol (Oxf). 2012 Oct;77(4):508-12. doi: 10.1111/j.1365-2265.2012.04450.x. PMID 22640465
- [Result] Hattersley JG, Pfeiffer AF, Roden M, Petzke KJ, Hoffmann D, Rudovich NN, Randeva HS, Vatish M, Osterhoff M, Goegebakan O, Hornemann S, Nowotny P, Machann J, Hierholzer J, von Loeffelholz C, Mohlig M, Arafat AM, Weickert MO. Modulation of amino acid metabolic signatures by supplemented isoenergetic diets differing in protein and cereal fiber content. J Clin Endocrinol Metab. 2014 Dec;99(12):E2599-609. doi: 10.1210/jc.2014-2302. PMID 25157543
- [Result] Cuthbertson DJ, Weickert MO, Lythgoe D, Sprung VS, Dobson R, Shoajee-Moradie F, Umpleby M, Pfeiffer AF, Thomas EL, Bell JD, Jones H, Kemp GJ. External validation of the fatty liver index and lipid accumulation product indices, using 1H-magnetic resonance spectroscopy, to identify hepatic steatosis in healthy controls and obese, insulin-resistant individuals. Eur J Endocrinol. 2014 Nov;171(5):561-9. doi: 10.1530/EJE-14-0112. PMID 25298375